CLINICAL TRIAL: NCT03944434
Title: Phase II, Multicenter, Single Arm Trial to Assess the Feasibility of First Line Ribociclib in Combination with a Non Steroidal Aromatase Inhibitor in Elderly Patients with Hormone Receptor Positive/HER2 Negative Advanced Breast Cancer
Brief Title: FACILE: FeAsibility of First-line RiboCIclib in OLdEr Patients with Advanced Breast Cancer
Acronym: FACILE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Sandro Pitigliani (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FACILE
Record Dates: First submitted 2019-04-09; First posted 2019-05-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: ribociclib; hormone receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Aromatase Inhibitors; Letrozole; Anastrozole; Gonadotropin-Releasing Hormone; Triptorelin Pamoate; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental): patients will receive anastrozole tablets (1 mg once daily) or letrozole tablets (2.5 mg once daily) + ribociclib tablets (600 mg day 1 to 21 in a 28 day cycle). Courses repeat every 28 days in the absence of disease progression, unacceptable toxicity, physician's decision, patient's refusal/consent withdrawal, or lost to follow-up.
  A LHRH agonist (triptorelin 3,75 mg or leuprolide 3,75 mg or goserelin 3,6 mg, as injectable intramuscular (i.m.) or subcutaneous (s.c.) implant every 28 days) will be used in men.
  Interventions: Drug: Ribociclib; Drug: Aromatase Inhibitors, non steroideal; Drug: LHRH agonist

INTERVENTIONS:
Drug: Ribociclib — ribociclib 600 mg/day orally
  Other Names: Kisqali
Drug: Aromatase Inhibitors, non steroideal — letrozole 2.5 mg/day orally or anastrozole 1 mg/day orally
  Other Names: Femara; Arimidex
Drug: LHRH agonist — Triptorelin 3,75 mg or Leuprolide 3,75 mg or goserelin 3,6 mg, as injectable.
  Other Names: Triptorelin; Leuprolide; Goserelin

SUMMARY:
Phase II, multicenter, single arm trial to assess the feasibility of first line ribociclib in combination with a non steroidal aromatase inhibitor in women or men aged 70 years-old or older, with hormone receptor positive/HER2 negative advanced breast cancer

DETAILED DESCRIPTION:
Elderly patients are generally more susceptible to the side effects of active treatments. Patients entered in clinical trials, especially the elderly, are not completely representative of the "real" population because of selection process. The lack of data collected from a real population turns the indication of treatment a challenging task and expose older patients to a risk of under treatment (fear of excessive toxicity because of the lack of data).

With the aim of covering this gap, we are planning to run a phase II trial evaluating the feasibility of delivering the combination of ribociclib plus NSAI as first-line treatment specifically in a population of breast cancer patients aged ≥70 years.

Primary endpoint:

• The treatment feasibility will be evaluated as the proportion of patients not having experienced disease progression (PD), still on treatment with ribociclib plus NSAI 6 months after the first drug administration

Secondary endpoints:

* Treatment adherence
* Safety and tolerability
* Patient reported outcomes (PROs)
* Overall response rate (ORR)
* Progression free survival (PFS)

ELIGIBILITY:
Inclusion Criteria:

1. Patients male or female, aged 70 years-old or older at the time of informed consent.
2. Patients with advanced (locoregionally recurrent or metastatic) breast cancer not amenable to curative therapy.
3. Measurable or not measurable but evaluable disease according to RECIST criteria 1.1
4. Patient has a histologically and/or cytologically confirmed diagnosis of estrogen receptor positive and/or progesterone receptor positive breast cancer by local laboratory.
5. Patient has a HER2 negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing.
6. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
7. Patient has an estimated life expectancy of > 24 weeks.
8. Patient has adequate bone marrow and organ function as defined by all of the following laboratory values (as assessed by local laboratory):

   1. Absolute neutrophil count ≥1.5 x 109/L
   2. Platelets ≥ 100 x 109/L
   3. Hemoglobin ≥ 9.0 g/dL
   4. Potassium, sodium, calcium corrected for serum albumin and magnesium within normal limits or corrected to within normal limits with supplements before first dose of the study medication
   5. INR ≤ 1.5
   6. Serum creatinine <1.5 mg/dl or creatinine clearance ≥50mL/min
   7. Total bilirubin < ULN except for patients with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN.
   8. In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be < 2.5 × ULN. If the patient has liver metastases, ALT and AST should be < 5 × ULN.
9. Patient must have a 12-lead ECG values with all of the following parameters at screening:

   1. QTcF interval at screening < 450 msec (using Fridericia's correction)
   2. Resting heart rate ≥50 bpm
10. Patient must be able to swallow ribociclib and NSAI tablets
11. Written informed consent must be obtained prior to any screening procedures
12. Patient must be able to communicate with the investigator and comply with the requirements of the study procedures.

Exclusion Criteria:

* 1. Patient has received prior treatment with chemotherapy or hormonal therapy (except for neoadjuvant/ adjuvant chemotherapy), or any CDK4/6 inhibitor.

NOTE:

* Patients who received (neo) adjuvant therapy for breast cancer are eligible. If the prior neo (adjuvant) therapy included letrozole or anastrozole the disease-free interval must be greater than 12 months from the completion of treatment until study entry.
* Patients who received ≤ 28 days of letrozole or anastrozole for advanced disease prior to inclusion in this trial are eligible.

  2. Patient has a known hypersensitivity to any of the excipients of ribociclib or NSAI 3. Patient in concurrently using other anti-cancer therapy. 4. Patient who has not had resolution of all acute toxic effects of prior anti-cancer therapy to NCI CTCAE version 5.0 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).

  5. Patient who has received extended-field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to start of treatment, and who has not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion). Patient from whom ≥ 25% of the bone marrow has been previously irradiated are also excluded 6. Patient has a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.

  7. Patient with central nervous system (CNS) metastases unless they meet all of the following criteria:
  1. At least 4 weeks from prior therapy for CNS disease completion (including radiation and/or surgery) to starting the study treatment.
  2. Clinically stable CNS lesions at the time of study treatment initiation and not receiving steroids and/or enzyme-inducing anti-epileptic medications for the management of brain metastases for at least 2 weeks.

     8. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., uncontrolled ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).

     9. Patient has a known history of HIV infection (testing not mandatory). 10. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgement, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g., chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.) 11. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

  <!-- -->

  1. History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
  2. History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  3. Documented cardiomyopathy
  4. Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block)
  5. Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

  i. Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia ii. Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (within 5 half-lives or 7 days prior to starting study drug) iii. Inability to determine the QTcF interval on screening f. Systolic Blood Pressure (SBP) >160 or <90 mmHg 12. Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug:
  1. Concomitant medications, herbal supplements, and/or fruits (e.g. grapefruit, pummeloes, star fruit, Seville oranges) and their juices that are strong inducers or inhibitors of CYP3A4/5,
  2. Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.

     13. Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment.

     NOTE:
* The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-11-27 (Estimated)

PRIMARY OUTCOMES:
Treatment feasibility | 6 months
  The treatment feasibility will be evaluated as the proportion of patients not having experienced disease progression (PD), still on treatment with ribociclib plus NSAI 6 months after the first drug administration

SECONDARY OUTCOMES:
Patient Diary | 36 months
  Diary to self-report data regarding taking medication and to evaluate treatment adherence
Incidence of Treatment-Emergent adverse events and serious adverse events (Safety and tolerability) | 36 months
  Adverse events (AE), AE of special interest and serious adverse events (SAE). CTCAE V. 5.0 will be adopted.
Patient reported outcomes (PROs) | 36 months
  PROs using Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire, score: 0= not at all; 1= a little bit; 2= somewhat; 3= quite a bit; 4= very much;
Overall response rate (ORR) | 36 months
  ORR as defined by RECIST 1.1 for patients with measurable disease
Progression free survival (PFS) | 36 months
  PFS as defined by RECIST 1.1 based on investigator' assessment
Number of comorbities (impact on study inclusion) | 30 months
  Number of comorbidities and relative grading will be collected using Cumulative Illness Rating Scale- Geriatric (CIRS-G) (for patients not included into the study due to comorbities).SCORE: 0- No problem , 1- Current mild problem or past significant problem, 2- Moderate disability or morbidity/requires first line therapy, 3- Severe/ constant significant disability/ uncontrollable chronic problems, 4- Extremely severe/ immediate treatment required/ end organ failure/ severe impairment in function

CONTACTS AND LOCATIONS:
Overall Officials: Laura Biganzoli, MD, Principal Investigator — Hospital of Prato
Locations (1):
- Hospital of Prato, Prato, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finn RS, Crown JP, Lang I, Boer K, Bondarenko IM, Kulyk SO, Ettl J, Patel R, Pinter T, Schmidt M, Shparyk Y, Thummala AR, Voytko NL, Fowst C, Huang X, Kim ST, Randolph S, Slamon DJ. The cyclin-dependent kinase 4/6 inhibitor palbociclib in combination with letrozole versus letrozole alone as first-line treatment of oestrogen receptor-positive, HER2-negative, advanced breast cancer (PALOMA-1/TRIO-18): a randomised phase 2 study. Lancet Oncol. 2015 Jan;16(1):25-35. doi: 10.1016/S1470-2045(14)71159-3. Epub 2014 Dec 16. PMID 25524798
- [Background] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- [Background] Hortobagyi GN, Stemmer SM, Burris HA, Yap YS, Sonke GS, Paluch-Shimon S, Campone M, Blackwell KL, Andre F, Winer EP, Janni W, Verma S, Conte P, Arteaga CL, Cameron DA, Petrakova K, Hart LL, Villanueva C, Chan A, Jakobsen E, Nusch A, Burdaeva O, Grischke EM, Alba E, Wist E, Marschner N, Favret AM, Yardley D, Bachelot T, Tseng LM, Blau S, Xuan F, Souami F, Miller M, Germa C, Hirawat S, O'Shaughnessy J. Ribociclib as First-Line Therapy for HR-Positive, Advanced Breast Cancer. N Engl J Med. 2016 Nov 3;375(18):1738-1748. doi: 10.1056/NEJMoa1609709. Epub 2016 Oct 7. PMID 27717303
- [Background] Goetz MP, Toi M, Campone M, Sohn J, Paluch-Shimon S, Huober J, Park IH, Tredan O, Chen SC, Manso L, Freedman OC, Garnica Jaliffe G, Forrester T, Frenzel M, Barriga S, Smith IC, Bourayou N, Di Leo A. MONARCH 3: Abemaciclib As Initial Therapy for Advanced Breast Cancer. J Clin Oncol. 2017 Nov 10;35(32):3638-3646. doi: 10.1200/JCO.2017.75.6155. Epub 2017 Oct 2. PMID 28968163
- [Background] Hortobagyi GN, Stemmer SM, Burris HA, Yap YS, Sonke GS, Paluch-Shimon S, Campone M, Petrakova K, Blackwell KL, Winer EP, Janni W, Verma S, Conte P, Arteaga CL, Cameron DA, Mondal S, Su F, Miller M, Elmeliegy M, Germa C, O'Shaughnessy J. Updated results from MONALEESA-2, a phase III trial of first-line ribociclib plus letrozole versus placebo plus letrozole in hormone receptor-positive, HER2-negative advanced breast cancer. Ann Oncol. 2018 Jul 1;29(7):1541-1547. doi: 10.1093/annonc/mdy155. PMID 29718092
- [Background] Rugo HS, Turner NC, Finn RS, Joy AA, Verma S, Harbeck N, Masuda N, Im SA, Huang X, Kim S, Sun W, Iyer S, Schnell P, Bartlett CH, Johnston S. Palbociclib plus endocrine therapy in older women with HR+/HER2- advanced breast cancer: a pooled analysis of randomised PALOMA clinical studies. Eur J Cancer. 2018 Sep;101:123-133. doi: 10.1016/j.ejca.2018.05.017. Epub 2018 Jul 25. PMID 30053671
- [Background] Sonke GS, Hart LL, Campone M, Erdkamp F, Janni W, Verma S, Villanueva C, Jakobsen E, Alba E, Wist E, Favret AM, Bachelot T, Hegg R, Wheatley-Price P, Souami F, Sutradhar S, Miller M, Germa C, Burris HA. Ribociclib with letrozole vs letrozole alone in elderly patients with hormone receptor-positive, HER2-negative breast cancer in the randomized MONALEESA-2 trial. Breast Cancer Res Treat. 2018 Feb;167(3):659-669. doi: 10.1007/s10549-017-4523-y. Epub 2017 Oct 22. PMID 29058175